CLINICAL TRIAL: NCT01135537
Title: Pharmacokinetics and Pharmacodynamics of Thymoglobulin in Paediatric Haematopoietic Stem-cell Transplant Recipients
Brief Title: Pharmacokinetics of Thymoglobulin in Paediatric Haematopoietic Stem-cell Transplants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed before 2017 due to inconclusive results from Lab
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Tal Schechter-Finkelstein, Staff Physician, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000013834
Record Dates: First submitted 2010-03-26; First posted 2010-06-02 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Malignancy; Metabolic Disease; Genetic Disorder
Keywords: allogeneic hematopoietic stem cell transplantation; pharmacokinetics; pediatrics
MeSH Terms: conditions — Neoplasms; Metabolic Diseases; Genetic Diseases, Inborn | interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thymoglobulin (Experimental): Thymoglobulin 7.5 mg/kg/course prior to HSCT
  Interventions: Biological: Thymoglobulin (rATG)

INTERVENTIONS:
Biological: Thymoglobulin (rATG) — Thymoglobulin 2.5 mg/kg of body weight IV administered daily for 3 days prior to HSCT.
  Thymoglobulin infused over a minimum of 6 hours for the first infusion and over at least 4 to 6 hours on subsequent days of therapy.
  Other Names: Anti-thymocyte Globulin (Rabbit)

SUMMARY:
This study will describe the pharmacokinetic disposition of biologically active rabbit anti-thymocyte globulin (rATG) after a consistent dose of 7.5 mg/kg/course given as part of the conditioning regimen in children undergoing hematopoeitic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Allogeneic hematopoeitic stem cell transplantation (HSCT) is a therapeutic option for patients with malignancies as well as metabolic and genetic diseases. Conditioning regimens given prior to donor cell infusion aim to ablate the recipient bone-marrow, to allow engraftment of the stem-cells infused, and to prevent acute versus host disease (aGVHD). Anti-thymocyte globulin (ATG) is one of the immunosuppressive drugs given as a preparative regimen for HSCT. Subjects will be given an ATG infusion daily for 3 days prior to HSCT and serum levels will be collected, as per schedule, with the last sample taken +100 days post-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled to receive ATG 2.5mg/kg/day for 3 days as part of the preparative regimen for HSCT, as determined by the responsible HSCT physician.
* Written, informed consent

Exclusion Criteria:

* Hypersensitivity to rabbit proteins or to any product excipients
* Active acute or chronic infections, which would contraindicate any additional immunosuppression
* Known pregnancy or breastfeeding

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Schechter-Finkelstein, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital For Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Related Info — http://doi.org/10.1016/j.bbmt.2011.12.258

RESULTS

PARTICIPANT FLOW:
Groups:
- Thymoglobulin: Thymoglobulin 7.5 mg/kg/course prior to HSCT
  Thymoglobulin (rATG): Thymoglobulin 2.5 mg/kg of body weight IV administered daily for 3 days prior to HSCT.
  Thymoglobulin infused over a minimum of 6 hours for the first infusion and over at least 4 to 6 hours on subsequent days of therapy.
Period: Overall Study
Arm/Group | Thymoglobulin
Started | 30
Completed | 17
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Disposition of ATG After a 7.5 mg/kg/Course
Description: ATG pharmacokinetic parameters were estimated using a noncompartmental model. Maximum Observed Concentration (Cmax) of ATG After a 7.5 mg/kg/Course was measured
Time Frame: 100 days
Population: Blood samples for ATG concentration determination were obtained at 0, +1, +4, +7, +14, +28, +60, +75 and +100 days post-HSCT. ATG serum concentrations were analyzed using a validated immunoassay. ATG pharmacokinetic parameters were estimated using a noncompartmental model. The relationship between HSCT outcomes
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 17
mg/L | 7.86 (2.9)

ADVERSE EVENTS:
Description: This is a pharmacokinetic study. There was no risk for the patients for measuring drug levels.
  Adverse Events were not monitored/assessed for this study.
Arm/Group | Thymoglobulin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes